CLINICAL TRIAL: NCT01236287
Title: Special Access for the Use of Voclosporin for Kidney Transplantation
Status: No longer available | Type: Expanded Access
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0904010380
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Immunosuppression; Transplantation, Kidney
MeSH Terms: interventions — voclosporin

INTERVENTIONS:
Drug: Voclosporin — Subjects will receive voclosporin capsules, twice daily

SUMMARY:
Voclosporin is an investigational medication previously studied to prevent acute rejection in patients who receive a kidney transplant. This study is a compassionate release program where subjects previously participating in the study entitled A Phase 2B, Randomized, Multicenter, Open-Label, Concentration Controlled, Safety Study of ISA247 and Tacrolimus (Prograf®) in denovo Renal Transplant Patients (ISA05-01)" may be eligible to continue to receive voclosporin despite the Phase 2B study being terminated by the sponsor. Under the compassionate release program, subjects previously taking voclosporin may continue to receive the study medication until the drug is FDA-approved and commercially available in the United States.

Voclosporin was approved by the FDA in January 2021 for the treatment of active lupus nephritis. The sponsor (now called Aurinia Pharma, U.S.) is willing to continue to provide voclosporin (commercial supply) for the one subject remaining in this special access protocol.

DETAILED DESCRIPTION:
Voclosporin is an investigational medication previously studied to prevent acute rejection in patients who receive a kidney transplant. This study is a compassionate release program where subjects previously participating in the study entitled A Phase 2B, Randomized, Multicenter, Open-Label, Concentration Controlled, Safety Study of ISA247 and Tacrolimus (Prograf®) in denovo Renal Transplant Patients (ISA05-01)" may be eligible to continue to receive voclosporin despite the Phase 2B study being terminated by the sponsor. Under the compassionate release program, subjects previously taking voclosporin may continue to receive the study medication until the drug is FDA-approved and commercially available in the United States.

Subjects will receive voclosporin and will be followed in an outpatient setting. After their initial visit, patients will return for follow-up at least every 3 months (through month 24) and then every 6 months (beginning at month 24). Safety and efficacy measurements will be taken at appropriate time points as outlined in the table below. Trough voclosporin measurements will be collected at least every 3 months (through month 24) and then every 6 months (beginning at month 24) or more frequently at clinic visits as appropriate (as indicated by clinical events (such as rejection, infection, adverse event) or concomitant administration of an interacting medication.

Starting at the month 144 visit, subjects sign an informed consent addendum, which describes the change to annual study visits moving forward. The subjects will continue to receive their current dose of voclosporin without therapeutic drug monitoring and will be followed in an outpatient setting. Patient and graft survival data will be collected on an annual basis for safety reporting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently enrolled in "A Phase 2B, Randomized, Multicenter, Open-Label, Concentration Controlled, Safety Study of ISA247 and Tacrolimus (Prograf®) in denovo Renal Transplant Patients (ISA05-01)" and has a compelling reason to remain on voclosporin
* Subjects must provide Informed Consent to participate in this study
* Females of child-bearing potential must have a negative pregnancy test prior to enrollment

Exclusion Criteria:

* Subjects who have already been switched off of voclosporin (ISA247) and on to another immunosuppressive agent

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Kapur, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/NewYork-Presbyterian Hospital, New York, New York, United States